CLINICAL TRIAL: NCT00572858
Title: Estrogen Deficiency and Cardiovascular Disease in Premenopausal Women
Status: Completed | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Noel Bairey Merz, Director, Cedars-Sinai Medical Center
Other Study IDs: IRB 6326
Record Dates: First submitted 2007-12-12; First posted 2007-12-13 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Estrogen Deficiency
Keywords: Hypo E
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood Hormone draw for FSH, E2; Urine Pregnancy test; Fasting lipid (cholesterol) panel, fasting insulin and fasting blood glucose levels; Reproductive hormones (FSH, LH, E1, E2, bioE2, PO, freeT, SHBG, DHEA-S); Plasma levels of inflammatory and endothelial function markers including but not limited to hsCRP, serum amyloid, endothelin-1, and ELAM; Fasting Salivary Cortisol (stress hormone).
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Premenopausal women: Female patients who have undergone coronary angiography and are under the age of 55
  Interventions: Procedure: Blood test; Genetic: Blood test; Procedure: Ultrasound of neck arteries; Procedure: Saliva test

INTERVENTIONS:
Procedure: Blood test — for cholesterol, glucose and insulin levels and levels of various hormones, including but not limited to estrogen
Genetic: Blood test — Blood test for genetic testing
Procedure: Ultrasound of neck arteries — Non-invasive test using ultrasound waves to measure the thickness of the arteries
Procedure: Saliva test — Saliva test for cotisol levels

SUMMARY:
For unexplained reasons, young premenopausal women with heart disease have twice the rate of death compared to men of the same age. Animal experiments have shown that stress can reduce ovary function in females monkeys due to reductions in brain hormones. This stress and reduced brain hormone levels lead to low estrogen levels and can cause menstrual cycles to become irregular, leading to reductions in fertility. These monkeys are also more likely to develop heart disease. In order, to better understand this relationship the investigators would like to study estrogen levels in premenopausal women with heart disease.

Premenopausal women who have recently undergone a study of their coronary (heart) arteries will have their blood hormone levels measured over one menstrual cycle. The investigators will correlate the blood hormone levels with coronary angiography results and with other markers of heart disease, such as a test that uses noninvasive, painless ultrasound waves to study the thickness of the arteries in the neck (carotid arteries). In addition blood cholesterol levels, blood sugar levels and other blood tests have been shown to correlate with heart disease will be measured.

Another aim of the study is to evaluate a potential link between environmental stress and hormone levels. Each patient will be given multiple questionnaires to evaluate stress, anxiety and depression and the investigators will be measuring the stress hormone (cortisol) levels in saliva for additional information.

The results of the study will further explore a possible link between low estrogen levels and heart disease in young premenopausal women and help pave the way for larger research studies to define better ways of preventing heart disease in these women.

DETAILED DESCRIPTION:
Specific Aims

1. To document that estrogen deficiency of hypothalamic (central brain) origin is a stable trait, when measured over one menstrual cycle or an approximate thirty days apart in premenopausal women undergoing angiography for coronary ischemia.
2. To document a relationship between estrogen deficiency, other reproductive hormones and environmental stress in premenopausal women.
3. To measure prevalence of angiographic coronary artery disease among premenopausal women and correlate it with noninvasive markers of coronary artery disease and the genetic relationship of estrogen in cardiovascular disease through genotyping and analysis of genes related to estrogen metabolism and pathways.

We are recruiting female patients who have undergone coronary angiography and are under the age of 55. After subject has signed the informed consent, we will screen her by testing her blood for two hormones to see if subject is premenopausal. If she is, she will be enrolled in the study and scheduled to return for a baseline visit on day 12-18 of the following menstrual cycle or 22-30 days later.

During the baseline visit we will measure height, weight, blood pressure, heart rate and waist-hip ratio. Subject will have to be fasting and we will draw blood for cholesterol, glucose and insulin levels and levels of various hormones, including but not limited to estrogen. Subject's saliva will be collected to test for cortisol levels. If subject agrees, a tablespoon of your blood will also be collected for genetic testing. Subject will be asked to fill out a separate consent form. Participation in the study does not mandate participation in genetic testing. Subject also will be given multiple questionnaires including questions regarding medical history, family history, medication use, stress, anxiety, and depression. They should be filled out within 48 hours of the blood draw to correlate findings. Neck arteries will be examined by ultrasound waves to measure the thickness of the arteries. This test can be performed on your second of third visit.

The final exit visit will be timed 26-33 days from your baseline visit. It will include all the tests that subjects underwent during their baseline visit except for the ultrasound, which will only be done once.

In summary, subjects will make three to four visits, the total study duration will be three to four months.

We will evaluate your hormone levels and other blood markers with respect to your coronary angiogram and thickness of the neck arteries. We will also assess whether your hormone levels are related to stress, anxiety and depression. And finally, we will measure the variability in your hormone levels over the testing period.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal by WISE criteria
* English speaking (for the purposes of complete psychosocial assessment)
* Able to give informed consent
* Clinically-indicated coronary angiography within the last 24 months prior to enrollment with no interim change in symptoms, hospitalization, or events.
* Non-English speaking patients will be consented but will not undergo psychosocial assessment as part of the study.

Exclusion Criteria:

* Pregnant or intention of becoming pregnant during study period.
* Current hormonal therapy (oral contraceptives, hormone replacement therapy, designer estrogens or phytoestrogens)
* History of bilateral salpingoophorectomy

Max Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Premenopausal Women
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2005-01; Primary Completion 2020-10 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
estrogen deficiency of hypothalamic (central brain) origin | 51 days
  at Baseline and Exit Visits (Baseline visit on day 12-18 of the following menstrual cycle; Final exit visit will be timed 26-33 days from the baseline visit).

CONTACTS AND LOCATIONS:
Overall Officials: C.Noel Bairey-Merz, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Women's Heart Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Demissie S, Cupples LA, Shearman AM, Gruenthal KM, Peter I, Schmid CH, Karas RH, Housman DE, Mendelsohn ME, Ordovas JM. Estrogen receptor-alpha variants are associated with lipoprotein size distribution and particle levels in women: the Framingham Heart Study. Atherosclerosis. 2006 Mar;185(1):210-8. doi: 10.1016/j.atherosclerosis.2005.06.008. Epub 2005 Jul 7. PMID 16005459
- [Background] Gold B, Kalush F, Bergeron J, Scott K, Mitra N, Wilson K, Ellis N, Huang H, Chen M, Lippert R, Halldorsson BV, Woodworth B, White T, Clark AG, Parl FF, Broder S, Dean M, Offit K. Estrogen receptor genotypes and haplotypes associated with breast cancer risk. Cancer Res. 2004 Dec 15;64(24):8891-900. doi: 10.1158/0008-5472.CAN-04-1256. PMID 15604249
- [Background] Herrington DM, Howard TD. ER-alpha variants and the cardiovascular effects of hormone replacement therapy. Pharmacogenomics. 2003 May;4(3):269-77. doi: 10.1517/phgs.4.3.269.22686. PMID 12718718
- [Background] Schuit SC, de Jong FH, Stolk L, Koek WN, van Meurs JB, Schoofs MW, Zillikens MC, Hofman A, van Leeuwen JP, Pols HA, Uitterlinden AG. Estrogen receptor alpha gene polymorphisms are associated with estradiol levels in postmenopausal women. Eur J Endocrinol. 2005 Aug;153(2):327-34. doi: 10.1530/eje.1.01973. PMID 16061840
- [Background] Schuit SC, Oei HH, Witteman JC, Geurts van Kessel CH, van Meurs JB, Nijhuis RL, van Leeuwen JP, de Jong FH, Zillikens MC, Hofman A, Pols HA, Uitterlinden AG. Estrogen receptor alpha gene polymorphisms and risk of myocardial infarction. JAMA. 2004 Jun 23;291(24):2969-77. doi: 10.1001/jama.291.24.2969. PMID 15213208
- [Background] Schuit SC, van der Klift M, Weel AE, de Laet CE, Burger H, Seeman E, Hofman A, Uitterlinden AG, van Leeuwen JP, Pols HA. Fracture incidence and association with bone mineral density in elderly men and women: the Rotterdam Study. Bone. 2004 Jan;34(1):195-202. doi: 10.1016/j.bone.2003.10.001. PMID 14751578
- [Background] Shearman AM, Cupples LA, Demissie S, Peter I, Schmid CH, Karas RH, Mendelsohn ME, Housman DE, Levy D. Association between estrogen receptor alpha gene variation and cardiovascular disease. JAMA. 2003 Nov 5;290(17):2263-70. doi: 10.1001/jama.290.17.2263. PMID 14600184
- [Background] Shearman AM, Demissie S, Cupples LA, Peter I, Schmid CH, Ordovas JM, Mendelsohn ME, Housman DE. Tobacco smoking, estrogen receptor alpha gene variation and small low density lipoprotein level. Hum Mol Genet. 2005 Aug 15;14(16):2405-13. doi: 10.1093/hmg/ddi242. Epub 2005 Jul 13. PMID 16014638